CLINICAL TRIAL: NCT01770600
Title: Assessment and Treatment of Impulsivity and Thought Process Disorder in Patients With Active Suicidal Ideation and Depression.
Brief Title: Impulsivity and Thought Process Disorder in Patients With Active Suicidal Ideation and Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never initiated, did different study
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Cheryl McCullumsmith, Division Director, Hospital Psychiatry, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F1003310002
Record Dates: First submitted 2012-08-07; First posted 2013-01-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Impulsivity; Active Suicidal Ideation; Depression
Keywords: Age 19 to 64; Medically stable; No current or history of psychosis; No alcohol or benzodiazepine withdrawal
MeSH Terms: conditions — Impulsive Behavior; Depression | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone (Active Comparator): Administer pill of risperidone 1 mg once a day by mouth for 5 days.
  Interventions: Drug: Riperidone
- Placebo (Placebo Comparator): Administer pill of placebo once a day by mouth for 5 days.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — placebo pill administered daily for 5 days
  Arms: Placebo
Drug: Riperidone — 1 mg risperidone administered orally for 5 days
  Other Names: risperdal
  Arms: Risperidone

SUMMARY:
This study is dedicated to achieving a better understanding of how the brain processes information. Specifically, the investigators are studying cognitive function, thought process, and impulsivity in people with and without suicidal thoughts. You are being asked to participate in a research study to learn how the use of a medication, risperidone, improves your symptoms of depression. Specifically the investigators are studying the effectiveness of reducing the thought of suicide and other symptoms of severe depression. Risperidone is approved by FDA for the treatment of schizophrenia and bipolar mania, and clinical practice suggests that it might benefit patients with major depressive disorder. During clinical trials with 2607 patients, risperidone was proved to be safe. This is a pilot study to test a new indication of risperidone for treatment of severe depression. The study medication will be given in addition to usual psychiatric care.

DETAILED DESCRIPTION:
Men and women between the ages of 19-64, who have a diagnosis of major depressive disorder, and are currently in a severe depressive episode with suicidal thoughts, are eligible to participate in this voluntary research study. A control group will consist of men and women between the ages of 19-64 who have a diagnosis or major depressive disorder and are currently in a severe depressive episode but are not having suicidal thoughts.

During the screening visit, appropriate demographic, medical, and psychiatric data will be collected, including a diagnostic assessment and an assessment of the severity of your depression. You will be asked to complete several pen and pencil questionnaires to learn more about your current state of mind. This evaluation will take approximately two hours. If you qualify for the control or assessment group, you will be asked to meet with researchers again at 2, 4 and 6 days after your initial evaluation. If you qualify for the study group, you will be randomly (like the flip of a coin) assigned by a computer to receive either risperidone (1-2 mg/day) or placebo once a day by mouth. You will take the study medication for 5 nights in addition to your standard of care antidepressant prescribed by your doctor.

Forty participants will enter a double-blind study, which means that neither you nor your doctors will know which study medicine (risperidone or placebo) you are receiving. If medically necessary, the medication information will be released so your doctor can find out what medicine you were randomly assigned to.

You will have a follow-up evaluation (either in the hospital or returning for an office visit) at Day 5. At this visit, you will be evaluated by a psychiatrist and will be asked to complete questionnaires designed to assess the effect of the study medications on your symptoms. At this visit you will also be asked about possible side effects and how you are tolerating the medicine. These visits should take approximately one hour each.

At the screening and the end of the five day treatment, additional neuropsychological evaluations will be administered to assess your progress. These additional assessments will take approximately one hour to complete.

Members of the control group will receive no study related medications and will not return for a follow up visit.

Information for Women of Childbearing Potential or Men Fathering a Child Because risperidone may affect mother's milk or a developing fetus, breast-feeding and pregnant women are not allowed to take part in the study. Women who can become pregnant must take a pregnancy test before the start of the study. Unless they cannot have children because of surgery or other medical reasons, men and women must have been using an effective method of birth control before starting the study. Effective birth control includes birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause pregnancy.

Optional functional MRI(fMRI) brain Sub-study

10 participants will participate in the fMRI sub-study, which will include a 5 day open-label trial of risperidone. An fMRI scan will be done prior to receiving study drug and 5 days later. During this fMRI, a picture of your brain will be obtained. The fMRI procedure requires you to lie still on a narrow table with a circular scanner around your head. The fMRI scan takes approximately 40 minutes. Two of the neuropsychological assessments will be administered during the scan. Sub-study participants will complete a computer-based version of the tasks that will be performed during the fMRI scan prior to the brain imaging session. This is necessary to ensure you understand the tasks you will be performing while the imaging is taking place. Electing not to participate in this sub-study will not jeopardize participation in the drug trial. A neurologist, Dr. Lawrence Ver Hoef will review the MRI scans for incidental findings.

ELIGIBILITY:
Inclusion Criteria:

* Age : 19-64
* Suicidality score of > 4 on Montgomery-Asberg Depression Rating Scale (MADRS)

Exclusion Criteria:

* pregnant,
* medically unstable,
* history of schizophrenia,
* schizoaffective disorder,
* bipolar disorder,
* psychosis NOS,
* urine drug screen positive for cocaine,
* marijuana or amphetamines,
* withdrawal from opiates,
* benzodiazepines or alcohol,
* currently on antipsychotic drug therapy. Also excluded are those subjects who require the use of mood stabilizers or antipsychotics.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Decrease in depression symptoms | baseline to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl B McCullumsmith, MD PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States